CLINICAL TRIAL: NCT03309176
Title: Is Endometrial Withdrawal Bleeding Necessary Prior to Ovulation Induction With Clomiphene Citrate? A Randomized Controlled Trial and Feasibility Study
Brief Title: "Stair Step Study"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL56254.091.15
Record Dates: First submitted 2017-08-09; First posted 2017-10-13 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-08

CONDITIONS: Ovulation Disorder
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: Stair step group: blind start ovulation induction (no progesterone induced withdrawal bleeding and stair step protocol in case of treatment failure.
  Control: standard care; a progesterone induced withdrawal bleeding in case of no spontaneous menses before starting an ovulation induction cycle and in between anovulatory cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): Intervention:Medroxyprogesterone acetate (Provera) 10 mg daily for 10 days will be used prior to starting ovulation induction with clomiphene citrate (CC) and between anovulatory cycles. On cycle day (CD) 3 CC 50 mg is administered daily for 5 days. Follicle growth will be monitored by ultrasound, starting from CD11. Anovulatory patients (defined as no follicle ≥ 14 mm) on CD20, will receive Provera 10mg daily for 10 days. The CC dosage will be increased in the next cycle. On CD3 patients will receive CC 100 mg daily for 5 days with ultrasounds performed from CD11 onwards. Anovulatory patients will receive Provera 10mg daily for 10 days. In the next cycle the CC dose will be increased to 150 mg, starting from CD3, daily for 5 days with ultrasounds starting from CD11-20.
  Interventions: Drug: Medroxyprogesterone Acetate 10 MG
- Stair Step group (Experimental): Intervention: Stair step protocol without medroxyprogesterone acetate 10 mg prior to ovulation induction with clomiphene citrate (CC), nor in between anovulatory cycles. After performing an ultrasound to check for the presence of cysts or any other abnormalities and a negative pregnancy test, patients will receive CC 50 mg daily for 5 days. Ultrasounds will be performed on CD11-14. If there is no response on CD14 (no follicle ≥ 14 mm), the dose of CC is immediately increased to 100 mg CC daily for 5 days and an ultrasound is performed 1 week following the last ultrasound. If there is no response, 150 mg CC daily is initiated immediately for 5 days and the ultrasound is repeated 1 week after the previous ultrasound.
  Interventions: Other: Stair step protocol without Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Medroxyprogesterone Acetate 10 MG — Patients in the standard arm will receive Medroxyprogesterone Acetate 10mg daily for 10 days prior to the first ovulation induction cycle and in between anovulatory cycles.
  Other Names: Provera
  Arms: Standard group
Other: Stair step protocol without Medroxyprogesterone Acetate — No administration of Medroxyprogesterone Acetate prior to each cycle. Stair step method: rapidly increasing the dose of clomiphene citrate in case of no follicular response
  Other Names: Stair step
  Arms: Stair Step group

SUMMARY:
Rationale:

There is some information suggesting that a progesterone-induced withdrawal bleeding before the start of ovulation induction in women suffering from oligo- or amenorrhea reduces pregnancy and live birth rate.

Objective:

To evaluate the effects of withholding progesterone-induced endometrial withdrawal bleeding before ovulation induction on the time to pregnancy and the ongoing pregnancy rate.

Study design:

Prospective multicenter randomized controlled feasibility study

Study population:

Women with oligomenorrhea or amenorrhea according to WHO classification category 2

Intervention:

Patients will be randomized to receive one of the following two treatments:

Stair step group: blind start ovulation induction (no progesterone induced withdrawal bleeding and stair step protocol in case of treatment failure.

Control: standard care; a progesterone induced withdrawal bleeding in case of no spontaneous menses before starting an ovulation induction cycle and in between anovulatory cycles.

Main study parameters/endpoints:

The primary endpoints are the time to pregnancy and ongoing pregnancy rate within a treatment horizon of 3 cycles. Secondary endpoints include time to ovulation, endometrial thickness, multiple pregnancy and the incidence of treatment failure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The number of site visits or physical examinations will not differ from accepted clinical practice.

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

To demonstrate whether withholding progesterone induced endometrial shedding prior to ovulation induction improves the ongoing pregnancy rate per cycle compared to not withholding progesterone treatment and to demonstrate its impact on the time to pregnancy.

Secondary objectives:

To elucidate the impact of the two study protocols on time to ovulation, endometrial thickness, multiple follicle growth, multiple pregnancy and the incidence of treatment failure. Furthermore, in accordance to the proposed areas of focus addressed by feasibility studies [Bowen et al (2009)], the number of eligible patients, the number of protocol violations and the number of drop-outs will be recorded.

STUDY DESIGN

Prospective multicenter randomized controlled study. The participating centers are:

* Radboud UMC, Nijmegen
* Canisius Wilhelmina Ziekenhuis (CWZ), Nijmegen
* Gelderse Vallei, Ede

Patients will be randomly allocated to receive one of the following treatment protocols:

* Standard group: medroxyprogesterone acetate (Provera®) 10 mg for 10 days prior to starting ovulation induction with CC and in between anovulatory cycles.
* Stair Step group: no Provera® prior to ovulation induction with CC, nor in between anovulatory cycles.

Standard group The standard group will receive our standard care. Provera® will be administered for 10 days (after a negative pregnancy test) to induce an endometrial whitdrawal bleeding. Menses may be expected as early as 3 days after the last pill. Prior to each treatment cycle, an ultrasound will be performed on cycle day 3 to check up on the presence of cysts after which CC 50 mg is administered for 5 days. Follicle growth will be monitored by ultrasound, starting from cycle day (CD) 11. If there is no response (defined as no follicle ≥ 14 mm) on CD 20, Provera® will be administered for 10 days. The CC dosage will be increased in the next cycle. Three days after the start of the next menses, patients will receive CC 100 mg for 5 days with follicle growth monitoring starting again from CD 11. Anovulatory patients (no follicle ≥ 14 mm) on CD 20 will receive Provera® for 10 days. Three days after the start of menses the CC dose will be increased to 150 mg and will be administered for 5 days with ultrasounds starting from CD 11-20.

Stair Step group The stair-step group will receive the following treatment: after performing an ultrasound to check for the presence of cysts or any other abnormalities and a negative pregnancy test, patients will be given CC 50 mg for 5 days. Ultrasounds will be performed on days 11-14. When there is no response on CD 14 (no follicle ≥ 14 mm), the dose of CC is immediately increased to 100 mg CC for 5 days and an ultrasound is performed 1 week following the last ultrasound. If there is no response, 150 mg CC is initiated immediately for 5 days and the ultrasound is repeated 1 week after the previous ultrasound.

In both arms, ovulation is confirmed by evidence of a preovulatory follicle followed by menses with onset at the expected time (cycle length of 25-35 days) or by pregnancy.The CC dose can be adjusted in case of a high response. Treatment failure is defined as failure to ovulate following CC 150 mg. Patients who conceive will receive an ultrasound examination at 8 weeks of gestation to confirm an ongoing pregnancy. Following this last scan the study period for the given patient will be completed. All patients will undergo a maximum of 3 treatment cycles as part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* WHO classification category 2 PCOS or non-PCOS
* Age between 18 - 41 years
* Patent Fallopian tubes, proven by hysterosalpingography (HSG), a negative Chlamydia antibody titre (CAT) or diagnostic laparoscopy combined with tubal testing (DLS and TT), depending on the local protocol.
* BMI < 40 kg/m2

Exclusion Criteria:

* BMI > 40 kg/m2
* Previous unsuccessful ovulation induction cycles with CC
* Double-sided tubal pathology
* Presence of ovarian cysts on ultrasound
* Moderate - severe male infertility (TMSC < 3 million)
* Grade III/IV endometriosis
* Thrombosis
* Severe liver disease

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate per cycle | in case of pregnancy: 8 weeks after the start of each cycle, (maximum of 3 cycles, duration of 1 cycle: 28-35 days)
  Ongoing pregnancy is defined as the presence of at least one intra uterine fetus with heartbeat at 8 weeks of gestation
Time to pregnancy | duration of 1 cycle: 28-35 days, a maximum of 3 cycles will be performed (pregnancy test will be performed at the end of the cycle if there is no menstruation)
  the time between obtaining informed consent and the presence of a positive pregnancy test after treatment

SECONDARY OUTCOMES:
Time to ovulation | 3 cycles of 28-35 days, calculated as 14 days before the start of menstruation or 14 days before a positive pregnancy test
  calculated as 14 days prior to the first day of menstruation or positive pregnancy test
Endometrial thickness on the last day of ultrasonography | maximum of 3 cycles (each 28-35 days)
  measurement of the endometrial thickness on the last day of ultrasound monitoring. This day can differ among cycles, depending on the speed of follicle growth, hence it cannot be further specified.
The incidence of multiple follicle growth on the last day of ultrasonography | maximum of 3 cycles (each 28-35 days)
  This day can differ among cycles, depending on the speed of follicle growth, hence it cannot be further specified.
The incidence of multiple pregnancy | in case of pregnancy: 8 weeks after the start of a treatment cycle (maximum of 3 cycles; each 28-35 days)
  ultrasound performed at 8 weeks of gestation, which is 8 weeks after the start of a treatment cycle
The incidence of treatment failure | maximum of 3 cycles (each 28-35 days)
  treatment failure is defined as no follicle ≥ 14 mm on CD 20 despite using a maximum clomiphene citrate dose of 150 mg in the standard arm. Or no follicle ≥ 14 mm after increasing the clomiphene citrate dose up to 150 mg.
The number of eligible patients | Inclusion 16 months, follow-up 3 months.
  The total number of patients that fits the inclusion criteria.
The number of protocol violations | duration: maximum of 3 cycles (each 28-35 days)
  The total number of protocol violations.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Gelderse Vallei Hospital, Ede, Gelderland
  - Canisius-Wilhelmina Hospital, Nijmegen, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No